CLINICAL TRIAL: NCT01250041
Title: Continuous Saphenous Block Vs. Continuous Femoral Block for Total Knee Arthroplasty: Prospective, Randomized, Double Blind Study.
Brief Title: Continuous Saphenous Block Versus Continuous Femoral Block for Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: JF Asenjo, MUHC
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 10-153-SDR
Record Dates: First submitted 2010-11-26; First posted 2010-11-30 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Total Knee Arthroplasty Secondary to Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- femoral block (Active Comparator)
  Interventions: Procedure: continuous femoral nerve block
- saphenous block (Experimental)
  Interventions: Procedure: continuous saphenous nerve block

INTERVENTIONS:
Procedure: continuous femoral nerve block — ultrasound guided femoral nerve catheter insertion.
  Arms: femoral block
Procedure: continuous saphenous nerve block — ultrasound guided saphenous nerve catheter insertion
  Arms: saphenous block

SUMMARY:
Strength of the Quadriceps Muscle is key to recover from Total Knee Arthroplasty. In this study we compare two techniques for pain control after total knee arthroplasty in terms of preserving the motor function (the strength of the quadriceps muscles of the thigh) which will facilitate the rehabilitation and accelerate the hospital discharge. We will use ultrasound guided technique to block either the femoral nerve in the control group or the saphenous nerve in the experimental group. The primary outcome is the functional capacity and the impact of each block on the ability to walk by measuring the distance patients are able to walk in two minutes in post operative day one in the two groups. The secondary outcome is the morphine consumption in the two groups.

ELIGIBILITY:
Inclusion Criteria:

- Subject age over 18 years coming for total knee arthroplasty secondary to osteoarthritis

Exclusion Criteria:

* ASA 4-5
* Abnormal liver enzymes, hepatic failure, renal failure and cardiac failure if they become contraindication for the use of regional anesthesia
* Contraindications for spinal anesthesia
* Morbid obesity
* Organ transplant
* Neuropathic pain
* History of stroke or major neurological deficit
* Sensory and motor disorders in the operated limb
* Previous drug dependency
* Chronic use of opioids
* Allergy to local anesthetics
* Inability to comprehend pain assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-08 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
to assess the functional capacity and the impact of each block on the ability to walk by measuring the distance (the 2 minute walk test) in post op day one in the two groups. | post op day one

SECONDARY OUTCOMES:
the morphine consumption in the two groups. | post op day one

CONTACTS AND LOCATIONS:
Overall Officials: JF Asenjo, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada